CLINICAL TRIAL: NCT01482676
Title: Investigating the Role of microRNAs in the Regulation of Gene Expression and Organ Remodeling During Lower Urinary Tract Dysfunction, Including Bladder Pain Syndrome/Interstitial Cystitis (BPS), and Overactive Bladder Syndrome (OAB)
Brief Title: The Role of microRNAs in Organ Remodeling in Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 146/05b
Record Dates: First submitted 2011-11-17; First posted 2011-11-30 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Prostatic Hyperplasia; Urinary Bladder Neck Obstruction; Cystitis, Interstitial
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neck Obstruction; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen cold-cut bladder biopsies preserved in RNAlater buffer or in SDS-PAGE sample buffer; PFA-fixed tissue, primary cultures of urothelium and smooth muscle
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: controls (normal bladder function)
- 2: acontractile bladder
- 3: overactive bladder
- 4: bladder pain syndrome

SUMMARY:
Urgency, frequency and incomplete emptying are the key symptoms of lower urinary tract dysfunction, including bladder pain syndrome/interstitial cystitis, and overactive bladder syndrome. Lower urinary tract dysfunction is associated with cellular stress, leading to changes in gene expression and consequent organ remodeling. MicroRNAs are small regulatory molecules, affecting protein synthesis. They are quickly winning recognition as potential therapeutic agents. The investigators will perform a comparative study of mRNAs changed in lower urinary tract dysfunction and address the role of differentially expressed miRNAs in regulation of the genes, important for bladder function. The experimental approach, combining the analysis of human biopsy material with the in vitro cell-based models, will allow the investigators to elucidate the effects of miRNAs on the expression of receptors, contractile proteins and tight junction proteins. Once the disease-induced miRNAs have been characterised and their target genes validated, it will be possible to influence their expression levels thus counter-acting their effects.

The investigators' work addresses fundamental mechanisms of signal transduction in urothelium and smooth muscle during cellular stress caused by inflammation or bladder outlet obstruction, and its regulation in the diseased state. The investigators' findings will further the knowledge of the molecular mechanisms of lower urinary tract dysfunction and have implications for diagnosis and treatment. Additionally, they have relevance for other clinical conditions, where miRNAs are implicated.

DETAILED DESCRIPTION:
Background

Urgency, frequency and incomplete emptying are the key symptoms of lower urinary tract (LUT) dysfunction, including bladder pain syndrome/interstitial cystitis (BPS), and overactive bladder syndrome (OAB). Detrusor overactivity, which causes the symptoms of overactive bladder syndrome, is commonly observed in patients with bladder outlet obstruction. LUT dysfunction is associated with cellular stress, characterised by changes in cell signalling and the consequent alterations of gene expression leading to organ remodelling. Previously the investigators showed that NK1R-mediated signalling was down-regulated in BPS patients, and implicated microRNAs (miRNAs) in the regulation of NK1R expression and function.

MicroRNAs (miRNAs) are quickly gaining recognition for their role in many biological processes and disease states. MiRNAs are endogenous non-coding single-stranded RNAs which regulate gene expression by post-transcriptional mechanisms. The microRNAs regulate thousands of human gene products, complicating the efforts to predict and functionally validate their targets. Since miRNAs are important for many basic biological processes, any deregulation in their biogenesis or function may develop into a medical condition. Here the investigators propose to investigate the role of miRNAs in gene regulation during LUT disorders.

Chronic BPS is a clinical syndrome characterised by urgency/frequency, pelvic pain and inflammation in the absence of a detectable agent. A multitude of pathogenetic mechanisms have been postulated, but an inflammatory component is commonly thought to be involved. Epithelial damage has often been invoked: the mucinous layer of the healthy bladder is often compromised in patients with BPS. An initiating event (toxin) may cause increased urothelial permeability, which in turn leads to nerve sensitisation. The resulting cell injury propagates, leading to a self-perpetuating inflammatory reaction.

Urgency is a pivotal symptom of the lower urinary tract, and also one of the most bothersome symptoms in men suffering from benign prostatic hyperplasia and the resulting bladder outlet obstruction (BOO). In women OAB is a dynamic disorder, and an estimated 34% of women above 40 experience significant urinary storage symptoms. In contrast to BPS, patients with overactivity do not report bladder pain, although the perception of urgency and the arising discomfort vary between individuals. In order to facilitate diagnosis of BPS and its distinction from DO, and offer specific treatment regimens for each disorder, it is important to unravel the mechanisms behind the pathophysiology of these diseases.

The investigators' previous results suggest that the diseased state of the human urinary bladder is concomitant with structural and functional changes in smooth muscle and urothelium. In obstructed bladders, the organ's adaptive response is often accompanied by replacement of smooth muscle contractile proteins with their non-muscle or embryonic isoforms. On the other hand, a continuous exposure to neurotransmitters and low pH during inflammation in BPS induces a significant down-regulation of the tachykinin receptors and tight junction proteins, which might be mediated by the up-regulated miRNAs.

The investigators propose to establish the individual gene expression patterns characteristic for BPS and overactive as well as acontractile bladders and determine the common mechanisms of the cellular stress responses. They will study the role of miRNAs in the regulation of receptor-mediated signalling, contractility and epithelial integrity in these LUT dysfunctions, and delineate the miRNA species, characteristic of each symptomatic complex. Based on this information, they will identify and functionally validate gene targets of miRNAs in urinary bladders in order to foster the development of customised therapies. By comparing the expression of regulatory miRNAs in overactive and acontractile bladders the investigators will delineate the factors influencing the switch between the two programmes. Using validated miRNA/mRNA target pairs in cell based models of urothelium and bladder smooth muscle, they will investigate how the persistent stress-induced signalling during disease affects the miRNA expression and function of their target proteins. The findings will extend the knowledge of the molecular mechanisms of LUT dysfunction and have implications for diagnosis and treatment of these disorders.

Patient selection and sample processing:

Four study groups will be defined according to the international guidelines and ICS terminology: controls, BPS, overactive and acontractile. Twenty clinically stable patients pro study group will be recruited based on the clinical findings (international prostate symptom score (IPSS), bladder diary over 48 h, O'Leary-Sant questionnaire and visual analogue scale for pain). Biopsies will be obtained in either general or spinal anesthesia transurethrally from the bladder dome with a biopsy tong. Biopsies will then be snap frozen in liquid nitrogen or submerged in RNAlater (Qiagen). All patients will be undergoing surgery independent of this study. Tissue from the bladder dome for primary cell cultures will be obtained from patients undergoing cystectomy or bladder augmentation for bladder dysfunction as a last therapeutic option after other less invasive therapeutic options have failed. Control tissue will be obtained from bladder cancer patients, who have no lower urinary tract symptoms aside from hematuria. RNA will be extracted, and the expression levels of selected genes analyzed using Taqman realtime PCR and gene expression arrays (Applied Biosystems). Calcium imaging will be used to monitor the receptor activation and protein levels analysed by SDS-PAGE and Western Blotting. Receptor tissue distribution will be analysed by immunocytochemistry.

Objective

To identify and functionally validate gene targets of miRNAs in urinary bladder in order to foster the development of customised therapies. By comparing the expression of regulatory miRNAs in overactive and acontractile bladders the investigators will delineate the factors influencing the switch between the two programmes. Using validated miRNA/mRNA target pairs in cell based models of urothelium and bladder smooth muscle, they will investigate how the persistent stress-induced signalling during disease affects the miRNA expression and function of their target proteins. The findings will extend the knowledge of the molecular mechanisms of LUT dysfunction and have implications for diagnosis and treatment of these disorders.

Methods

RNA will be extracted, and the expression levels of selected genes analyzed using Taqman realtime PCR and gene expression arrays (Applied Biosystems). Calcium imaging will be used to monitor the receptor activation and protein levels analysed by SDS-PAGE and Western Blotting. Receptor tissue distribution will be analysed by immunocytochemistry.

ELIGIBILITY:
Inclusion Criteria:

* prostate hyperplasia
* bladder acontractility
* bladder pain
* age over 18 years old
* willingness to participate (informed concent)

Exclusion Criteria

* Age ≤ 18 years old
* Pregnancy
* History of or current genito-urinary tuberculosis
* History of pelvic surgery in the last 6 months
* History of bladder malignancy, high grade dysplasia or carcinoma in situ
* sexually transmitted diseases (STD's)
* Bacteriuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Department of Urology, Inselspital Bern, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Molecular traits of bladder dysfunction | 3 years

SECONDARY OUTCOMES:
MiRNA expression profiling of individual groups | 3 years
Protein expression profiling of individual groups | 3 years
Functional differences between groups | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Katia Monastyrskaya, PhD, Principal Investigator — Department of Urology, Bern University hospital
Locations (1):
- Department of Urology, Bern University hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Bartel DP. MicroRNAs: target recognition and regulatory functions. Cell. 2009 Jan 23;136(2):215-33. doi: 10.1016/j.cell.2009.01.002. PMID 19167326
- [Background] Cardozo LD, Van Kerrebroeck PE, Staskin DR. Considerations for the management of urgency symptoms in patients with overactive bladder syndrome. World J Urol. 2009 Dec;27(6):755-63. doi: 10.1007/s00345-009-0455-4. PMID 19690868
- [Background] Donaldson MM, Thompson JR, Matthews RJ, Dallosso HM, McGrother CW; Leicestershire MRC Incontinence Study Group. The natural history of overactive bladder and stress urinary incontinence in older women in the community: a 3-year prospective cohort study. Neurourol Urodyn. 2006;25(7):709-16. doi: 10.1002/nau.20235. PMID 16998862
- [Background] Keay S. Cell signaling in interstitial cystitis/painful bladder syndrome. Cell Signal. 2008 Dec;20(12):2174-9. doi: 10.1016/j.cellsig.2008.06.004. Epub 2008 Jun 19. PMID 18602988